# Prism Adaptation in Left Brain Stroke NCT04387162 02/07/22

#### Consent to be a Research Subject

## You Are Being Asked to Be in a Research Study

Concise presentation of key concepts

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study, you will be one of 100 people who are being studied at the Atlanta VA Health Care System.

#### Why is this study being done?

This study is being done to answer the question: Can we adapt spatial, motor and pain assessments and treatment procedures for people with aphasia and memory impairment? You are being asked to be in this research study because you are 18-89 years old and have aphasia and memory impairment caused by stroke.

#### Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care for your condition. Before you make your decision, you should take time to learn about the study.

#### What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will participate in up to 18 study visits lasting 1-3 hours each. The researchers will ask you to do the following:

- 8 assessment sessions (before treatment, during treatment, after treatment)
- 10 sessions of spatial retraining treatment (5 days per week for 2 weeks)

#### How is this study going to help you?

If you are in the study, you will be helping the researchers answer the study question. You will also receive information about your language, memory, spatial, and motor function, functional abilities and pain. You will also receive 10 sessions of spatial retraining treatment.

#### What are the risks or discomforts I should know about before making a decision?

The study will take time. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious. For this study, these include frustration or anxiety, nausea, loss of privacy, and breach of confidentiality. A full list of expected risks, their frequency and severity are in the RISKS section of this document. A full list of expected risks, their frequency and severity are in the RISKS section of this document.

#### **Alternatives to Joining This Study**

You do not have to be in this study to receive treatment. The study investigator can discuss alternative treatment options that may be available if you want this information.

#### What Should I Do Next?

Read this form, or have it read to you. Make sure the study doctor or study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.) Take time to consider this and talk about it with your family and friends.

**TITLE:** Prism Adaptation and Left Brain Stroke Rehabilitation

PRINCIPAL INVESTIGATOR: Amy Rodriguez, PhD

**SPONSOR'S NAME**: Department of Veterans Affairs

#### **PURPOSE**:

You are being asked to volunteer in a research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any benefits. If you decide not to take part in this study, your doctor will continue to treat you.

#### Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form, you will not give up any legal rights.

The purpose of the study is to investigate adapted methods for assessing and treating spatial and motor function and pain in patients with aphasia and memory impairment.

#### **CLINICALTRIALS.GOV:**

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that can identify you. At most the Web site will include a summary of the results. You can search this website at any time.

#### WHAT WILL I BE ASKED TO DO?:

You will be asked to take part in a study that includes up to 18 sessions that include assessment and/or treatment. The assessments will happen weekly for 8 weeks (8 sessions). Within the 8 weeks, you will receive treatment for 2 weeks. The treatment schedule will be 5 days per week during those 2 weeks (10 sessions). Each study visit will last approximately 1-3 hours. All visits will take place either by audio (phone) or video conference or face-to-face at the Atlanta VA Health Care System at 1670 Clairmont Rd. Decatur, GA 30033.

#### Assessment Sessions (8 sessions)

We will conduct assessments of your language, memory, spatial and motor abilities as well as your overall functioning. We will also ask you to complete questionnaires about pain. Some will be paper and pencil tests, and some will require you to answer questions or complete tasks in person or on a computer. We may audio or video record your responses. The recordings, used to score the tests, will be obtained for research purposes only. The recordings will not be disclosed outside of the VA. A research assistant will be with you at all times. You may request rest breaks between tests, and you may stop at any time. If you have participated in Dr. Rodriguez's study entitled "Intention Treatment for Anomia" (IRB#116056), we may obtain your data on certain cognitive and language assessments. We will only share data from these assessments to decrease testing burden. All other assessment data will be collected only for this research study and will not be shared as outlined in confidentiality section. Assessments will be conducted before the treatment program begins, during the treatment program, and after the treatment program ends. Some participants will have two testing sessions before the start of treatment, one testing session during treatment and five testing sessions after treatment. Some participants will have four testing sessions before the start of treatment, one session during treatment and three testing sessions after treatment. We are testing the how the assessments we administer should be adapted for participants with aphasia and memory impairment, and the assessments will help us measure the effect of treatment.



#### Prism Adaptation Treatment (10 sessions)

Prism Adaption Treatment (PAT) will be administered 5 days per week for 2 weeks (10 sessions) by a trained study clinician. PAT is a spatial retraining approach that involves repeated arm movements to visual targets while wearing goggles that shift the visual field horizontally. The goggles create a prismatic distortion that makes it appear that objects in the environment are displaced to the left. With the goggles on, reaching movements are shifted to the left of a fixed target. Over repeated attempts, the fixed target is reached. After removing the goggles, visual information returns to normal, but the spatial-motor system is more likely to direct movement to the right. We are testing the how PAT needs to be adapted

for participants with aphasia and memory impairment and the impacts of increased movement into the neglected (right) space.

#### Table of Study Activities

| Study Visit | Activity | # of<br>sessions | # of hours<br>per<br>session |
|---|---|---|---|
| Assessment<br>(before, during,<br>after treatment) | Before treatment: Language, memory, spatial, motor, pain, and functional ability tests | Up to 8 | 1-3 |
| | During treatment: Spatial, motor, pain, and functional ability tests | | |
| | After treatment: Spatial, motor, pain, and functional ability tests | | |
| Treatment | Prism Adaptation Treatment<br>Nausea profile (first three days) | 10 | <u>&lt;</u> 1 |

#### RISKS:

There may be side effects from the study device or procedures that are not known at this time.

#### Testing and treatment:

You may experience some frustration during testing of language, memory, spatial or motor functions. You may also feel frustrated during treatment. This frustration is tolerated well by most participants. If you become frustrated, you can ask to take a break to allow the frustration to go away. You may also experience nausea wearing the goggles. During the first three treatment sessions, we will use a questionnaire to find out if you are experiencing nausea. We will discontinue the treatment if nausea continues.

As with all research, there is a chance that confidentiality could be compromised; however, we take precautions to minimize this risk.

Participation in more than one research study may further increase risks to you. If you are already enrolled in another research study, please inform Amy Rodriguez (404-321-6111 x204201) or the person reviewing this consent before you enroll in this or any other research study.

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

#### **BENEFITS:**

Taking part in this research study may not benefit you personally. However, you will receive information about your language, memory, spatial, motor function, functional abilities and pain. You will also receive 10 sessions of spatial retraining. This research study may help us better understand how to adapt assessments and treatments for people with aphasia and memory impairment. It will also help us understand the impact of treatment, which can be used to help other people in the future.

#### **COMPENSATION:**

You will not pay for any of the study tests or procedures. Participants are compensated up to \$270 for completing the study. This compensation includes \$15 for each of the 18 study visits. Payments will be disbursed once all study visits are completed or at the time of withdraw or termination.

You will get emergency medical care if you get injured from being in this study. Under Federal Law, you will qualify for follow-up treatment if the injury was related to the research study. You may or may not get further compensation if you are injured in this study. This rule would not apply if you do not follow study procedures. If you believe you have been injured by this research, you should contact Amy Rodriguez, PhD at 404-321-6111 x204201.

#### COSTS:

You will not be charged for any treatments or procedures that are part of this study. However, some Veterans are required to pay co-payments for medical care and services provided by the VA. These co-payment requirements will continue to apply to medical care and services that are not part of this study.

You will get necessary medical treatment if you get injured from being in this study. This requirement does not apply to:

- (1) Treatment for injuries due to non-compliance by a subject with study procedures; or
- (2) Research conducted for VA under a contract with an individual or a non-VA institution.

If you believe you have been injured by this research, you should contact Amy Rodriguez at 404-321-6111 x204201

#### **ALTERNATIVES:**

You do not have to be in this study to receive treatment. The study investigator can discuss alternative treatment options that may be available if you want this information.

#### **HOW WILL MY PRIVATE INFORMATION BE PROTECTED:**

We will keep information about you, including any research records we create, strictly confidential to the extent required by law.

We may be required to release your record if we receive a subpoena or a court order. The study staff will keep your study files locked in a file cabinet in a private office. We will use a study number rather than your name on study records when we can. Your name and other facts that might point to you will not appear when we present this study or publish its results. People other than those doing this research study may have access to your medical and study records including:

- Department of Veterans Affairs
- The Office for Human Research Protections
- The Government Accountability Office (GAO)
- The Office of Research Oversight (ORO)
- The Inspector General
- Emory University
- Any appropriate state or federal government agencies that make rules and policy about how research is done that are not listed above
- IRB 116056

All research records and/or identifiers will be destroyed in accordance with the VA record retention schedule.

If you are a veteran who is a patient at the Atlanta VA Health Care System, a copy of your signed and dated consent and HIPAA forms may be placed in your medical record(s). If you are a <u>non-veteran</u> receiving clinical services (i.e., use of the laboratory, radiology, audiology, etc.) as part of this study, you will have an electronic medical record created for you. You will also be given a VA Notice of Privacy Practices (NOPP) and we will ask you to sign a form saying that you have received this notice.

If you are participating in a study where a test and/or procedure may be performed at Emory and you are not and have never been an Emory patient, you do not have an electronic medical record. Please note that an Emory medical record will be created if you have any services or procedures done by an Emory provider or facility for this study.

#### **HEALTH INFORMATION PORTABILITY AND ACCOUNTABILITY ACT (HIPAA):**

There are rules to protect your private health information. Federal and state laws and the federal medical law, known as the HIPAA Privacy Rule, also protect your privacy. By signing this form, you provide your permission called your 'authorization,' for the use and disclosure of information protected by the HIPAA Privacy Rule.

The research team working on the study will collect information about you. This includes things learned from the procedures described in this consent form. They may also collect other information including your name, address, date of birth, and information from your medical records such as diagnoses, progress notes, lab or radiology findings.

The research team may also need to disclose your health information and the information it collects to others as part of the study progress. Others may include the Office of Human Research Protections (OHRP), the VA Office of Research Oversight (ORO), and the Government Accountability (GAO), Emory University and the Emory Institutional Review Board, and Food and Drug Administration (FDA).

Your health information disclosed pursuant to this authorization may no longer be protected by Federal laws or regulations and may be subject to re-disclosure by the recipient.

You can revoke this authorization, in writing, at any time. To revoke your authorization, you must write to the Release of Information Office at this facility or you can ask a member of the research team to give you a form to revoke the authorization. Your request will be valid when the Release of Information Office receives it. If you revoke this authorization, you will not be able to continue to participate in the study. This will not affect your rights as a VHA patient to treatment or benefit outside of the study.

If you revoke this authorization, Amy Rodriguez (PI) and her research team can continue to use information about you that was collected before receipt of the revocation. The research team will not collect information about you after you revoke the authorization.

Treatment, payment or enrollment/eligibility for benefits cannot be conditioned on you signing this authorization. This authorization will expire at the end of the research study unless revoked prior to that time.

#### **RESULTS:**

Upon request, the study team can give you copies of your test scores without any clinical interpretation.

#### **CONFLICT OF INTEREST: None**

#### **IDENTIFIABLE PRIVATE INFORMATION**

Identifiers might be removed from the identifiable private information or identifiable biospecimens that are collected. After that removal, the information or biospecimens could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative

#### **CONTACT PERSONS:**

If you have any questions, concerns, or complaints about this study you can call a member of the study staff: Amy Rodriguez at 404-321-6111 x204201.

If you have been harmed from being in this study call: Amy Rodriguez at 404-321-6111 x204201.

If you want to speak to someone who is not a member of the study to discuss problems, ask questions or voice concerns, you can call:

The Research Compliance Officer at (404) 321-6111 ext. 206964 or the Clinical Studies Center Manager at (404) 321-6111 ext. 206933.

If you have any questions about your rights as a participant in this research study, call the Emory University Institutional Review Board at (404) 712-0720 or toll free at 1-877-503-9797.

#### **VOLUNTARY PARTICIPATION AND WITHDRAWAL:**

The study doctors have the right to end your participation in this study for any of the following reasons: If it would be dangerous for you to continue, if you do not follow study procedures as directed by the study doctors, or if the sponsor decides to end the study.

Your participation is voluntary and you have the right to refuse to be in this study. You can stop at any time after giving your consent. This decision will not affect in any way your current or future medical care or any other benefits to which you are otherwise entitled. For your safety, however, you should consider the study doctor's advice about how to go off the study treatment.

The study doctor, investigator, or sponsor may stop you from taking part in this study at any time if they decide it is in your best interest or if you do not follow study instructions.

We will give you a copy of this consent form to keep. If you are willing to volunteer for this research, please sign below.



### **RESEARCH PARTICIPANT'S SIGNATURE AND DATE:**

| Research Participant's name (Print) | |
|-------------------------------------|------|
| Decemb Destiningst's Cignoture | Data |
| Research Participant's Signature | Date |